CLINICAL TRIAL: NCT03976063
Title: Tocolysis in the Management of Preterm Premature Rupture of Membranes Before 34 Weeks of Gestation: a Double-blinded Randomized Controlled Trial
Brief Title: Tocolysis in the Management of Preterm Premature Rupture of Membranes Before 34 Weeks of Gestation
Acronym: TOCOPROM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Ministry of Health, France (Other Government); Groupe de Recherche en Obstétrique et Gynécologie (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P160917
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Preterm Premature Rupture of Membrane
Keywords: Preterm premature rupture of membranes; Tocolysis; Nifedipine; Latency; Neonatal outcome; Preterm birth; Randomized controlled trial
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Premature Birth | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nifedipine (Active Comparator)
  Interventions: Drug: Nifedipine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of Nifedipine

INTERVENTIONS:
Drug: Nifedipine — Loading dose: Oral Nifedipine 20 mg prolonged-release at T0 and T0.5 (i.e. 30 min), total=2x20 mg Maintenance dose: Oral Nifedipine 20 mg prolonged-release at T3, then 1 pill every 8 hr for 48 hr (i.e. T11, T19, T27, T35 and T43, total=6x20 mg)
  Arms: Nifedipine
Drug: Placebo of Nifedipine — Oral Placebo of Nifedipine 20 mg, at T0, T0.5, T3, T11, T19, T27, T35 and T43
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether short-term (48 hr) tocolysis reduces perinatal morti-morbidity in cases of PPROM at 22 to 33 completed weeks' gestation.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) complicates 3% of pregnancies and accounts for one-third of preterm births. It is a leading cause of neonatal mortality and morbidity and increases the risk of maternal infectious morbidity. In cases of early PPROM (22 to 33 completed weeks' gestation), expectant management is recommended in the absence of labor, chorioamnionitis or fetal distress. Antenatal steroids and antibiotics administration are recommended by international guidelines. However, there is no recommendation regarding tocolysis administration in the setting of PPROM. In theory, reducing uterine contractility should delay delivery and reduce risks of prematurity and neonatal adverse consequences. Likewise, a prolongation of gestation may allow administering a corticosteroids complete course that is associated with a two-fold reduction of morbidity and mortality. However, tocolysis may prolong fetal exposure to inflammation and be associated with higher risk of materno-fetal infection, potentially associated with neonatal death or long-term sequelae, including cerebral palsy.

The purpose of this study is to assess whether short-term (48 hr) tocolysis reduces perinatal morti-morbidity in cases of PPROM at 22 to 33 completed weeks' gestation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm premature rupture of membranes (PPROM) between 220/7 - 336/7 weeks of gestation, as diagnosed by obstetric team
* Singleton gestation
* Fetus alive at the time of randomization (reassuring fetal heart monitoring)
* 18 years of age or older
* French speaking
* Affiliated to social security regime or an equivalent system
* Informed consent and signed

Exclusion Criteria:

* PPROM ≥ 24 hours before diagnosis
* Ongoing tocolytic treatment at the time of PPROM
* Tocolytic treatment with Nifedipine between PPROM diagnosis and randomization
* Fetal condition contraindicating expectant management including chorioamnionitis, placental abruption, intrauterine fetal demise, non-reassuring fetal heart rate at the time of randomization
* Cervical dilation > 5 cm
* Iatrogenic rupture caused by amniocentesis or trophoblast biopsy
* Major fetal anomaly
* Maternal allergy or contra-indication to Nifedipine or placebo drug components*:

  * Myocardial infarction
  * Unstable angina pectoris
  * Hepatic insufficiency
  * Cardiovascular shock
  * Beta blockers

placebo drug components: lactose monohydrate, colloidal silica, microcrystalline cellulose

* Coadministration of diltiazem or rifampicin
* Hypotension (systolic pressure < 90 mmHg)
* Participation to another interventional research (category 1) in which intervention could interfere with TOCOPROM's results (efficacy and safety)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Perinatal morti-morbidity | Up to discharge from hospital, with a maximum of 24 weeks after birth.
  Composite outcome including fetal death, neonatal death and/or neonatal severe morbidity (mechanical ventilation ≥ 48 hrs, severe bronchopulmonary dysplasia, severe intraventricular hemorrhage, cystic periventricular leucomalacia, neonatal early-onset sepsis, necrotizing enterocolitis, retinopathy of prematurity).

SECONDARY OUTCOMES:
Prolongation of gestation | Up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Latency duration (defined as the duration from PPROM to delivery)
Prolongation of gestation | Up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Pregnancy prolongation beyond 48 hours after randomization
Prolongation of gestation | Up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Pregnancy prolongation beyond 1 week after randomization
Prolongation of gestation | Up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Gestational age at delivery
Prolongation of gestation | Up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Delivery after 37 weeks of gestation
Maternal morbidity | During the first 10 days postpartum
  Endometritis, based on clinical diagnosis associating fever (temperature ≥ 38.0°C) with uterine tenderness, purulent or foul-smelling lochia, and in the absence of any other cause.
Maternal morbidity | At delivery
  Intra-uterine infection, defined as fever (maternal temperature ≥38 °C), with no alternative cause identified, associated with at least two of the following criteria: persistent fetal tachycardia > 160 bpm, uterine pain or painful uterine contractions or spontaneous labor, purulent amniotic fluid.
Fetal mortality | Up to delivery so up to 20 weeks after PPROM (i.e. up to the maximum duration of a normal pregnancy)
  Fetal death
Neonatal mortality | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Neonatal death
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Mechanical ventilation ≥ 48 hrs
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Severe bronchopulmonary dysplasia
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Severe intraventricular hemorrhage
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Cystic periventricular leucomalacia
Neonatal severe morbidity | From birth to Day 3 after birth.
  Early-onset sepsis
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Necrotizing enterocolitis
Neonatal severe morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Retinopathy of prematurity
Neonatal morbidity | At birth.
  Severe fetal acidemia
Neonatal morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Respiratory distress syndrome
Neonatal morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Mild or moderate bronchopulmonary dysplasia
Neonatal morbidity | From birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Grades I-II intraventricular hemorrhage
Neonatal morbidity | From Day 3 after birth to discharge from hospital, with a maximum of 24 weeks after birth.
  Late-onset sepsis.
Vital status | At 22-26 months of corrected age
  Death between discharge and follow up at 2 years
Frequency of Gross motor impairment among children alive at 2 years of corrected age | At 22-26 months of corrected age
  Cerebral palsy
Frequency of Neurosensory impairment among children alive at 2 years of corrected age | At 22-26 months of corrected age
  Visual impairment
Frequency of Neurosensory impairment among children alive at 2 years of corrected age | At 22-26 months of corrected age
  Hearing impairment

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Kayem, MD, PhD, Principal Investigator — INSERM UMR 1153, Obstetrical, Perinatal and PEdiatric Epidemiology (EPOPé) Research Team, Center of Research in Epidemiology and Statistics Sorbonne Paris Cité (CRESS), DHU Risks in Pregnancy, Paris Descartes University, Trousseau University Hospital; Elsa Lorthe, RM, PhD, Study Director — INSERM UMR 1153, Obstetrical, Perinatal and PEdiatric Epidemiology (EPOPé) Research Team, Center of Research in Epidemiology and Statistics Sorbonne Paris Cité (CRESS), DHU Risks in Pregnancy, Paris Descartes University
Locations (1):
- Trousseau University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mackeen AD, Seibel-Seamon J, Muhammad J, Baxter JK, Berghella V. Tocolytics for preterm premature rupture of membranes. Cochrane Database Syst Rev. 2014 Feb 27;2014(2):CD007062. doi: 10.1002/14651858.CD007062.pub3. PMID 24578236
- [Background] Lorthe E, Goffinet F, Marret S, Vayssiere C, Flamant C, Quere M, Benhammou V, Ancel PY, Kayem G. Tocolysis after preterm premature rupture of membranes and neonatal outcome: a propensity-score analysis. Am J Obstet Gynecol. 2017 Aug;217(2):212.e1-212.e12. doi: 10.1016/j.ajog.2017.04.015. Epub 2017 Apr 13. PMID 28412086
- [Background] Couteau C, Haumonte JB, Bretelle F, Capelle M, D'Ercole C. [Management of preterm and prelabour rupture of membranes in France]. J Gynecol Obstet Biol Reprod (Paris). 2013 Feb;42(1):21-8. doi: 10.1016/j.jgyn.2012.10.008. Epub 2012 Nov 24. French. PMID 23182704
- [Background] Schmitz T, Sentilhes L, Lorthe E, Gallot D, Madar H, Doret-Dion M, Beucher G, Charlier C, Cazanave C, Delorme P, Garabedian C, Azria E, Tessier V, Senat MV, Kayem G. Preterm premature rupture of the membranes: Guidelines for clinical practice from the French College of Gynaecologists and Obstetricians (CNGOF). Eur J Obstet Gynecol Reprod Biol. 2019 May;236:1-6. doi: 10.1016/j.ejogrb.2019.02.021. Epub 2019 Mar 2. PMID 30870741
- [Background] Flenady V, Wojcieszek AM, Papatsonis DN, Stock OM, Murray L, Jardine LA, Carbonne B. Calcium channel blockers for inhibiting preterm labour and birth. Cochrane Database Syst Rev. 2014 Jun 5;2014(6):CD002255. doi: 10.1002/14651858.CD002255.pub2. PMID 24901312
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- [Derived] Lorthe E, Kayem G; TOCOPROM Study Group and the GROG (Groupe de Recherche en Obstetrique et Gynecologie). Tocolysis in the management of preterm prelabor rupture of membranes at 22-33 weeks of gestation: study protocol for a multicenter, double-blind, randomized controlled trial comparing nifedipine with placebo (TOCOPROM). BMC Pregnancy Childbirth. 2021 Sep 8;21(1):614. doi: 10.1186/s12884-021-04047-2. PMID 34496799